CLINICAL TRIAL: NCT02351908
Title: A Phase IV, Open-label Three-arm Study Investigating the Impact of a Combination of Tenofovir Disoproxil Fumarate/Emtricitabine With Raltegravir or Dolutegravir or Elvitegravir/Cobicistat on Renal Tubular Function and Renal Transporters in HIV-1 Antiretroviral naïve Patients
Brief Title: Renal Integrase Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SSAT 066
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-04

CONDITIONS: HIV
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; elvitegravir; Cobicistat; Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Racivir; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Stribild® (Tenofovir Disoproxil Fumarate, Elvitegravir, Cobicistat150mg/150mg/200mg/245mg) tablet 1 once daily for 48 weeks
  Interventions: Drug: Stribild® (Tenofovir Disoproxil Fumarate, Elvitegravir, Cobicistat)
- Arm 2 (Experimental): Isentress® (Raltegravir 400 mg) 1 tablet twice a day + Truvada® (FTC & Tenofovir) 1 tablet once a day for 48 weeks
  Interventions: Drug: Isentress® (Raltegravir 400 mg)1 tablet twice a day + Truvada® (FTC & Tenofovir) 1 tablet
- Arm 3 (Experimental): Tivicay® (Dolutegravir 50 mg) 1 tablet once a day + Truvada® (FTC & Tenofovir) 1 tablet once a day for 48 weeks
  Interventions: Drug: Tivicay® (Dolutegravir 50 mg) 1 tablet once a day + Truvada® (FTC & Tenofovir)

INTERVENTIONS:
Drug: Stribild® (Tenofovir Disoproxil Fumarate, Elvitegravir, Cobicistat)
  Arms: Arm 1
Drug: Isentress® (Raltegravir 400 mg)1 tablet twice a day + Truvada® (FTC & Tenofovir) 1 tablet
  Arms: Arm 2
Drug: Tivicay® (Dolutegravir 50 mg) 1 tablet once a day + Truvada® (FTC & Tenofovir)
  Arms: Arm 3

SUMMARY:
The purpose of this study is to observe the safety of Truvada® (TDF/FTC) in relation to its impact on kidney function combined with different Integrase Inhibitors (Dolutegravir, or Elvitegravir/Cobicistat or Raltegravir), when given to patients who are commencing treatment for HIV infection for the first time.

All three combinations (Raltegravir + Truvada®, Dolutegravir + Truvada® and Stribild®, a single pill which contains Elvitegravir/Cobicistat/Truvada®) are currently recommended by the national guide-lines and used in standard clinical practice.

DETAILED DESCRIPTION:
The study will monitor kidney function, and compare the safety and effectiveness of Truvada® when taken with Dolutegravir, or Elvitegravir/Cobicistat or Raltegravir, over the first 48 weeks of treatment in HIV-1 antiretrovirals naïve patients.

The safety and how well these drug combinations are tolerated will be determined based on physical examinations, laboratory tests, and questions about any problems the participant might experience during the study. As part of this trial, levels of HIV-1 in the blood and urinary markers of kidney function and inflammatory markers will be measured at various times during the study.

The total duration of participant involvement in the trial will be up to 48 weeks, with up to 45 days between the screening and baseline visits. Participants will need to visit the clinic 6 times within the 48 weeks.

Once participants have been confirmed to be eligible to participate in the study, participants will attend for a baseline visit (day 1) where they will be randomly assigned to receive one of the three treatments listed below:

* Treatment Arm 1: Stribild® (EVG/COBI/FTC/TDF) 1 tablet once a day
* Treatment Arm 2: Isentress® (Raltegravir 400 mg) 1 tablet twice a day + Truvada® 1 tablet once a day
* Treatment Arm 3: Tivicay® (Dolutegravir 50 mg) 1 tablet once a day + Truvada® 1 tablet once a day

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female aged 18 years or above
2. Has documented HIV-1 infection
3. Has signed the Informed Consent Form voluntarily
4. Is willing to comply with the protocol requirements, including dosing schedules of each regimen
5. Has a HIV-plasma viral load at screening >1000 copies/mL
6. Has any CD4 cell count
7. Has never been exposed to ART (other than via PEP or PREP, not associated with acquisition of HIV)
8. Has an estimated glomerular filtration rate (MDRD method) >60 ml/min
9. Has no known resistance to TDF and FTC or to Integrase Inhibitors. HIV resistance test has to be dated no more than 1 year prior screening date. Only a RT/Pr gene resistance test is re-quired.
10. If female and of childbearing potential, she is using effective birth control methods (as agreed by the investigator) and is willing to continue practising these birth control methods during the trial and for at least 30 days after the end of the trial (or after last intake of investigational ARVs); Dosing of the OCP may need to be adjusted if randomized to the Stribild® arm.

    Note: Women who are postmenopausal for least 2 years, women with total hysterectomy, and women who have a tubal ligation are considered of non-childbearing potential
11. If a heterosexually active male, he is using effective birth control methods and is willing to con-tinue practising these birth control methods during the trial and until follow-up visit

Exclusion Criteria:

1. Is infected with HIV-2
2. Is using any concomitant therapy disallowed as per SPC for the study drugs
3. Has a currently active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV Infection-1993) with the following exceptions (must be discussed with the sponsor prior to enrolment):

   * Stable cutaneous Kaposi's Sarcoma (no pulmonary or gastrointestinal involvement other than oral lesions) unlikely to require systemic therapy during the trial period
   * CD4 count less than 200 cells/mm3 Note: Primary and secondary prophylaxis for an AIDS defining illness is allowed
4. Has diabetes or any known or established renal disease or abnormality regardless of if stable
5. Has presence at screening of proteinurea and or a urinary protein/creatinine ratio >30
6. Has untreated / not well controlled hypertension
7. Has acute viral hepatitis including, but not limited to, A, B, or C
8. Has chronic hepatitis B or chronic hepatitis C with AST and/or ALT >5 x ULN Note: Subjects co-infected with chronic HCV (but not B) can enter the trial if clinically stable and not expected to require treatment during the trial period.
9. Has received any investigational drug within 30 days prior to the trial drug administration
10. No baseline resistance test to reverse transcriptase inhibitors available
11. Clinically significant allergy or hypersensitivity or other contraindication to any trial medication or excipients
12. If female, she is pregnant or breastfeeding
13. Screening blood results with any grade 3 / 4 toxicity according to Division of AIDS (DAIDS) grading scale, except: asymptomatic grade 3 glucose, amylase or lipid elevation or asymptomatic grade 4 triglyceride elevation (re-test allowed).
14. Clinical or laboratory evidence of significantly decreased hepatic function or decompensation: INR > 1.5 or albumin < 30g/L
15. Any condition (including drug/alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the trial.
16. Is not using high protein training supplements such as creatinine or intermittently following exclusionary or high protein diets
17. Is not receiving medication with known relevant drug interactions or contraindications to any of the trial medications

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in retinol-binding protein/creatinine ratio (PCR) with each regimen over 24 weeks. | 24 weeks
  The change in retinol-binding protein/creatinine ratio (PCR) with each regimen over 24 weeks (measured via nephelometric assay run on Siemens BNII nephelometer).

SECONDARY OUTCOMES:
Change in retinol-binding protein/creatinine ratio with each regimen over 12 and 48 weeks. | 48 weeks
  The change in retinol-binding protein/creatinine ratio (PCR) with each regimen over 12 and 48 weeks (measured via nephelometric assay run on Siemens BNII nephelometer)
eGFR | 48 weeks
  The variation from baseline of eGFR (C-G, MDRD with creatinine, CKD-EPI with creatinine / cystatin-C), creatinine, β2- and alpha1- microglobulin excretion, urinary albumin and pro-tein/creatinine ratio, urinary cystatin-C / creatinine ratio, fractional phosphate excretion (fasted plasma PO4 and urinary spot phosphate), plasma urate and rates of normoglycemic glycosuria on each regimen at week 4, 12, 24, 36, and 48 of therapy.
Virologic response | 48 weeks
  The proportion of patients achieving virologic response (HIV RNA < 40 cp/mL) on each regimen at week 4, 12, 24, 36 and 48.
Immunologic markers | 48 weeks
  The changes in immunologic markers (CD4+, CD8+, ratio) at weeks 4, 12, 24, 36 and 48 of therapy with each regimen.
Inflammatory markers | 48 weeks
  The changes in inflammatory markers (hsCRP, IL-6, d-dimer) at weeks 4, 12, 24 and 48 of therapy with each regimen.
Metabolic markers | 48 weeks
  The changes, from baseline in metabolic markers: lipids (TC, LDL, HDL, TGs), at 4, 12, 24, 36 and 48 weeks of therapy, and in insulin, fasting glucose and HOMA-i at 24 weeks of therapy with each regimen.
Tenofovir concentration | 4 weeks
  To measure tenofovir concentration (Ctrough 12 or 24) in plasma and urine, at week 4 of treat-ment with each regimen.
Genetic polymorphisms | 48 weeks
  Relationship between genetic polymorphisms and exposure to the studied drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Moyle, MD, MBBS, Dip GUN, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- SSAT Clinical Research Facility, London, United Kingdom